CLINICAL TRIAL: NCT03494933
Title: Re-evaluation of Optimal Re-synchronisation Therapy in Patients With Chronic Heart Failure - An Investigator-initiated, Event-driven, Prospective, Parallel-group, Randomised, Open, Blinded Outcome Assessment (PROBE), Multi-centre Trial Without Investigational Medical Products (Proof of Strategy Trial)
Brief Title: Re-evaluation of Optimal Re-synchronisation Therapy in Patients With Chronic Heart Failure
Acronym: RESET-CRT
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: End of the Funding period, no further funding to complete the trial could be saved
Sponsor: Helios Health Institute GmbH (Other)
Collaborators: Heart Center Leipzig - University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HRC048864
Record Dates: First submitted 2018-03-15; First posted 2018-04-11 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2022-08

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CRT-P group (Experimental): Intervention: CRT-P implantation
  Interventions: Procedure: CRT-P implantation
- CRT-D group (Active Comparator): Intervention: CRT-D implantation
  Interventions: Procedure: CRT-D implantation

INTERVENTIONS:
Procedure: CRT-P implantation — Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure and will receive on top a CRT-P device.
  Arms: CRT-P group
Procedure: CRT-D implantation — Patients will be treated according to Optimal Medical Therapy defined by ESC Guidelines for treatment of patients with heart failure and will receive on top a CRT-D device.
  Arms: CRT-D group

SUMMARY:
The objective of the study is to demonstrate that in patients with chronic heart failure who receive optimal medical treatment for this condition and have indication for Cardiac Resynchronisation Therapy, the implantation of a pacemaker (index group) is not inferior to defibrillator (control group) with respect to all-cause mortality.

DETAILED DESCRIPTION:
Heart failure is a leading cause of death, hospitalisation, impaired quality of life and health expenditure. Symptoms and survival can be significantly improved by implantation of a device for Cardiac Resynchronisation Therapy (CRT). CRT devices are available as biventricular pacemakers (CRT-P) or as significantly more complex and cost-intensive biventricular defibrillators (CRT-D).

In patients who have previously experienced a life-threatening arrhythmia, the choice of the CRT-D (and not the CRT-P) is imperative but these are a small minority of patients. For the vast majority of patients receiving CRT therapy, there is currently considerable uncertainty as to whether the defibrillator function is needed and whether its benefits outweigh its risks. The defibrillator function may protect patients from sudden cardiac death. On the other hand, device-associated complications such as device infections appear to be increased; furthermore the defibrillator comes along with specific adverse events, particularly inappropriate shocks. These shocks are common and not only traumatic to patients (potentially leading to post-traumatic stress syndrome, anxiety disorders and depression), they also are negatively associated with overall survival.

The objective of the trial is to demonstrate that in patients with chronic heart failure who receive optimal medical treatment for this condition and have indication for CRT, the implantation of a CRT-P (index group) is not inferior to CRT-D (control group) with respect to all-cause mortality. Patients with an indication for CRT will be randomised to CRT-P or CRT-D.

RESET-CRT is an event-driven trial with a planned number of randomised and treated patients of at least n=1,356 (maximum of 2,004) and of 361 primary endpoints within an estimated median follow-up period of about 29 to 40 months.

No investigational medical product is defined to be used within RESET-CRT since only the therapeutic strategy (CRT-D versus CRT-P) is a pre-defined study treatment and allocated by random group (Proof of Strategy Trial). The devices to be implanted will be decided by the treating physician on the basis of the situation of the individual study patient and in line with local policies in routine clinical care.

Duration of study period:

Enrolment of 1,356 patients is expected to be completed within 52 months after inclusion of the first patient, i.e., by 31 December 2022. With an overall annual event rate between 9.0% and 12.5%, 361 primary endpoints will have occurred within 9 to 20 months of randomisation of the last patient (between 30 September 2023 and 31 August 2024). Under these circumstances, the total study duration will be between 62 and 73 months.

The Steering Committee of the study might prolong the recruitment period, for instance by 12 months, in the event of an unexpected slower recruitment rate or an overall event rate < 9.0% for the primary endpoint.

For individual patients, the expected median follow-up time is between 29 and 40 months, with a minimum between 9 and 20 months and a maximum between 61 and 72 months. Follow-up may be prolonged by 12 months in the event of a prolonged recruitment period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years.
* Symptomatic chronic heart failure due to ischemic or non-ischemic cardiomyopathy with NYHA class II, III or ambulatory IV.
* Reduced left ventricular ejection fraction ≤35% in transthoracic echocardiography (TTE) or cardiac magnetic resonance imaging (MRI) assessed verifiably within 4 weeks prior to or on the day of enrolment.
* On Optimal Medical Therapy (OMT) for at least 3 months prior to enrolment.
* Class I or IIa indication for implantation of a device for cardiac resynchronisation therapy (according to 2016 Guidelines of the European Society of Cardiology for the diagnosis and treatment of acute and chronic heart failure).
* Signed informed consent.

Exclusion criteria:

* Class I or IIa indication for implantation of an ICD for secondary prevention of sudden cardiac death and ventricular tachycardia (according to the 2015 Guidelines of the European Society of Cardiology for the management of patients with ven-tricular arrhythmias and the prevention of sudden cardiac death).
* Violation of Instruction For Use of the selected device by at least one of the random group treatments.
* Ventricular tachycardia induced in an electrophysiological study.
* Carrying any implanted cardiac pacemaker, defibrillator or CRT device.
* Unexplained syncope.
* Hospitalised with unstable heart failure with NYHA class IV within 1 month prior to enrolment.
* Acute coronary syndrome or cardiac revascularization therapy by coronary angioplasty or coronary artery bypass grafting within 6 weeks prior to enrolment.
* Cardiac valve surgery or percutaneous cardiac valvular intervention such as transcatheter aortic valve replacement or transcatheter mitral valve repair performed within 3 months prior to enrolment.
* Reversible non-ischemic cardiomyopathy such as acute viral myocarditis or discontinuation of alcohol in alcohol-induced heart disease.
* On the waiting list for heart transplant.
* Any disease that limits life expectancy to less than 2 years.
* Severe chronic renal disease (GFR<15 ml/min and/or the need for dialysis)
* Participation in another clinical trial, either within the past 3 months or still ongoing (participation in sub-studies connected to this trial and participation in observational studies permitted).
* Previous participation in RESET-CRT.
* Pregnant women or women of childbearing potential not on adequate birth control.
* Drug abuse or clinically manifest alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-02-21 (Actual)

PRIMARY OUTCOMES:
Time from randomisation to the occurrence of all-cause death | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Time from randomisation to the occurrence of all-cause death

SECONDARY OUTCOMES:
Time from randomisation to death from cardiac causes | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Time from randomisation to death from cardiac causes
Time from randomisation to sudden cardiac death | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Time from randomisation to sudden cardiac death
Time from randomisation to life-threatening arrhythmias | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Time from randomisation to life-threatening arrhythmias
Time from randomisation to first composite of Major Adverse Cardiac Event (MACE) | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Time from randomisation to first composite of Major Adverse Cardiac Event (MACE)
Time from randomisation to first hospitalisation for cardiovascular reasons | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Time from randomisation to first hospitalisation for cardiovascular reasons
Nights spent in hospital for cardiovascular reasons per year of follow-up | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Number of nights spent in hospital is calculated as time difference in days from hospital discharge to hospital admission. All hospital stays are serious adverse event by definition and will be assessed by an independent Endpoint Review Committee. The Endpoint Review Committee will also evaluate if a hospital stay for cardiovascular reasons is given. Per year of follow-up refers to a calculated number related to total follow-up duration of each patient normalised to years of follow-up.
Number of hospital readmissions for cardiovascular reasons after randomisation | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  Number of hospital readmissions for cardiovascular reasons after randomisation
Changes in quality of life (EQ-5D) comparing inclusion/enrolment with 12 and 24 months | at baseline, 12 and 24 months after randomisation
  Quality of life will be measured using the European Quality of life 5 Dimension (EQ5D) questionnaire including its visual-analogue scale (Scores range from 0-100 where 0 is the worst score).
Total cost of treatment as compound endpoint of MACEs, number of hospital days for cardiovascular reasons and ambulatory visits for cardiovascular reasons | Randomization to end of study (event-driven, expected about 9 to 20 months after last patient in)
  otal cost of treatment as compound endpoint of MACEs, number of hospital days for cardiovascular reasons and ambulatory visits for cardiovascular reasons

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Hindricks, MD, Principal Investigator — Heart Center Leipzig - University Hospital
Locations (113):
- Germany (113):
  - Helios Klinikum Aue, Aue
  - Zentralklinik Bad Berka, Bad Berka
  - Universitäts-Herzzentrum, Bad Krozingen
  - Marienhaus Klinikum im Kreis Ahrweiler, Bad Neuenahr-Ahrweiler
  - RHÖN-KLINIKUM Campus Bad Neustadt, Bad Neustadt A.d. Saale
  - Herz- und Diabeteszentrum NRW - Universitätsklinik der Ruhr-Universität Bochum, Bad Oeynhausen
  - Segeberger Kliniken, Bad Segeberg
  - Maria-Hilf-Krankenhaus Bergheim, Bergheim
  - Sana Klinikum Lichtenberg, Berlin
  - Unfallkrankenhaus Berlin, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Jüdisches Krankenhaus Berlin, Berlin
  - Charité Campus Virchow-Klinikum, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Immanuel Klinikum Bernau - Herzzentrum Brandenburg, Bernau bei Berlin
  - Klinikum Bielefeld, Bielefeld
  - Berufsgenossenschaftliches Universitätsklinikum Bergmannsheil, Bochum
  - Augusta Kliniken Bochum, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Knappschaftskrankenhaus Bottrop, Bottrop
  - REGIOMED-KLINIKEN Klinikum Coburg, Coburg
  - St. Vinzenz-Hospital, Cologne
  - Herzzentrum Uniklinik Köln, Cologne
  - Krankenhaus Porz am Rhein, Cologne
  - Carl-Thiem-Klinikum, Cottbus
  - Helios Amper-Klinikum Dachau, Dachau
  - Klinikum Lippe Detmold, Detmold
  - St.-Johannes-Hospital Dortmund, Dortmund
  - Herz Zentrum Westfalen - Knappschaftskrankenhaus Dortmund, Dortmund
  - Praxisklinik Herz und Gefäße, Dresden
  - Herzzentrum Dresden Universitätsklinik, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - Hermann-Josef-Krankenhaus Erkelenz, Erkelenz
  - Universitätsklinikum Erlangen, Erlangen
  - Contilia Herz- und Gefäßzentrum, Essen
  - Ev.-Luth. Diakonissenanstalt zu Flensburg, Flensburg
  - Universitätsklinikum Frankfurt, Frankfurt am Main
  - Kreiskrankenhaus Freiberg, Freiberg
  - Klinikum Fulda, Fulda
  - UKGM - Universitätsklinikum Gießen, Giessen
  - Asklepios Harzklinik Goslar, Goslar
  - Helios Klinikum Gotha, Gotha
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Klinikum Gütersloh gGmbH, Gütersloh
  - Evangelisches Krankenhaus Hagen-Haspe, Hagen
  - Krankenhaus Martha-Maria Halle-Dölau, Halle
  - Universitätsklinikum Halle (Saale), Halle
  - Universitätsklinikum Hamburg-Eppendorf (UKE), Hamburg
  - Asklepios Kliniken Hamburg GmbH - Asklepios Klinikum Harburg, Hamburg
  - Asklepios Kliniken Hamburg GmbH, Hamburg
  - Albertinen Herz- und Gefäßzentrum - Albertinen Krankenhaus, Hamburg
  - St. Marien-Hospital Hamm, Hamm
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Helios St. Marienberg Klinik Helmstedt, Helmstedt
  - Oberhavel Kliniken, Hennigsdorf
  - Helios Klinikum Hildesheim, Hildesheim
  - Universitätsklinikum des Saarlandes, Homburg
  - Klinikum Ingolstadt, Ingolstadt
  - Universitätsklinikum Jena, Jena
  - Westpfalz-Klinikum GmbH, Kaiserslautern
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - B. Braun Ambulantes Herzzentrum Kassel, Kassel
  - Universitätsklinikum Schleswig-Holstein Campus Kiel, Kiel
  - Städtisches Krankenhaus Kiel, Kiel
  - Katholisches Klinikum Koblenz - Montabaur, Koblenz
  - Helios Klinikum Krefeld, Krefeld
  - Universitätsklinikum Leipzig, Leipzig
  - Herzzentrum Leipzig, Leipzig
  - Klinikum Leverkusen, Leverkusen
  - Cardio Centrum Ludwigburg, Ludwigsburg
  - Universitätsklinikum Schleswig-Holstein, Lübeck
  - Klinikum Lüdenscheid, Lüdenscheid
  - St.-Marien-Hospital Lünen, Lünen
  - Universitätsklinikum Magdeburg, Magdeburg
  - Johannes Wesling Klinikum Minden, Minden
  - Ev. Krankenhaus Bethesda Mönchengladbach, Mönchengladbach
  - Kliniken Maria Hilf, Mönchengladbach
  - Städtische Kliniken Mönchengladbach - Elisabeth-Krankenhaus Rheydt, Mönchengladbach
  - Klinik Augustinum, München
  - LMU Klinikum, München
  - Technische Universität München, München
  - München Klinik Neuperlach, München
  - Universitätsklinikum Münster, Münster
  - Havelland Kliniken, Nauen
  - Marienhaus Klinikum St. Elisabeth Neuwied, Neuwied
  - Klinikum Nürnberg Süd, Nuremberg
  - St. Vincenz-Krankenhaus, Paderborn
  - Helios Vogtland-Klinikum Plauen, Plauen
  - Harzklinikum Dorothea Christiane Erxleben Klinikum Quedlinburg, Quedlinburg
  - Elblandklinikum Riesa, Riesa
  - Universitätsmedizin Rostock, Rostock
  - Asklepios Klinikum Uckermark, Schwedt
  - Helios Kliniken Schwerin, Schwerin
  - Helios Klinikum Siegburg, Siegburg
  - Marien Kliniken, Siegen
  - Diakonie Klinikum Jung-Stilling, Siegen
  - Krankenhaus Maria-Hilf Stadtlohn Klinikum Westmünsterland, Stadtlohn
  - Johanniter-Krankenhaus Genthin-Stendal, Stendal
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Klinikum Landkreis Tuttlingen, Tuttlingen
  - Universitätsklinikum Ulm, Ulm
  - Aller-Weser-Klinik - Krankenhaus Verden, Verden an der Aller
  - Schwarzwald-Baar Klinikum, Villingen-Schwenningen
  - Helios Klinikum Warburg GmbH, Warburg
  - Sophien- und Hufeland-Klinikum, Weimar
  - Rems-Murr-Klinikum Winnenden, Winnenden
  - Helios Universitätsklinikum Wuppertal, Wuppertal
  - Universitätsklinikum Würzburg, Würzburg
  - Heinrich-Braun-Klinikum, Zwickau

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chatterjee NA, Poole JE. Cardiac Resynchronization Therapy in Nonischemic Cardiomyopathy: To D or P? JACC Heart Fail. 2021 Jun;9(6):450-452. doi: 10.1016/j.jchf.2021.04.001. Epub 2021 May 12. No abstract available. PMID 33992569